CLINICAL TRIAL: NCT00431782
Title: An Open-Label Multi-Center Study of ATI-5923 for Anticoagulation in Patients With Atrial Fibrillation
Brief Title: Study of a New Anticoagulant Drug in Patients With Atrial Fibrillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ARYx Therapeutics (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATI-5923-CLN-504
Record Dates: First submitted 2007-02-02; First posted 2007-02-06 (Estimated); Last update posted 2007-11-08 (Estimated); Status verified 2007-05

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Anticoagulation
MeSH Terms: conditions — Atrial Fibrillation | interventions — tecarfarin

INTERVENTIONS:
Drug: ATI-5923

SUMMARY:
The primary purpose of this study (CLN-504) is to determine the safety and develop a dosing regimen of an investigational anticoagulant drug (ATI-5923) in patients with atrial fibrillation.

DETAILED DESCRIPTION:
ATI-5923 is a structural analog of warfarin that is being developed as an oral anticoagulant. It has a similar pharmacological profile to warfarin but was designed to provide more uniform and stable anticoagulation. ATI-5923 is a selective, non-competitive inhibitor of vitamin K epoxide reductase. ATI-5923 is metabolized by esterase to a single inactive metabolite and thus is expected to have less variable metabolism, drug-drug interactions and reduced instances of under/over coagulation, making the response safer and more predictable. The primary purpose of this study is to develop a dosing regimen and INR monitoring schedule that can be applied in an outpatient setting to safely and conveniently anticoagulate patients with atrial fibrillation to a therapeutic INR. Patients with atrial fibrillation (AF) were chosen for the study population of this trial because they require anticoagulation if they have risk factors for stroke.

ELIGIBILITY:
Inclusion Criteria:

* Documented atrial fibrillation
* Candidate for anticoagulation or currently receiving warfarin at screening
* Males or females greater than 18 years of age
* Males or females with a CHADS2 score of 0 to 2

Exclusion Criteria:

* Contraindications to anticoagulation e.g., active bleeding
* Taking other anticoagulant or antiplatelet agents other than low-dose aspirin
* History of myocardial infarction, acute coronary syndrome, or coronary revascularization procedure within the past 3 months prior to Day 1
* History of laboratory values suggestive of anemia (i.e., Hb <10 gm/dL)
* Women of childbearing potential

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-12; Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
INR, Coagulation Factors II, VII, IX and X. Safety Measures: ECG, Laboratory and Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Dave Ellis, M.D., Ph.D, Study Director — ARYx Therapeutics
Locations (11):
- United States (11):
  - ARYx Investigational Site, Anaheim, California
  - ARYx Investigational Site, Yuba City, California
  - ARYx Investigational Site, Deerfield Beach, Florida
  - ARYx Investigational Site, Winfield, Illinois
  - ARYx Investigational Site, Oklahoma City, Oklahoma
  - ARYx Investigational Site, Wellsboro, Pennsylvania
  - ARYx Investigational Site, Wynnewood, Pennsylvania
  - ARYx Investigational Site, Greer, South Carolina
  - ARYx Investigational Site, Spartanburg, South Carolina
  - ARYx Investigational Site, Memphis, Tennessee
  - ARYx Investigational Site, San Antonio, Texas

REFERENCES:
- [Derived] Ellis DJ, Usman MH, Milner PG, Canafax DM, Ezekowitz MD. The first evaluation of a novel vitamin K antagonist, tecarfarin (ATI-5923), in patients with atrial fibrillation. Circulation. 2009 Sep 22;120(12):1029-35, 2 p following 1035. doi: 10.1161/CIRCULATIONAHA.109.856120. Epub 2009 Sep 8. PMID 19738136